CLINICAL TRIAL: NCT02210065
Title: The Pre-Emptive Use of Recipient-Derived Autologous Cytomegalovirus (CMV)-Specific Cytotoxic T Cells for Cytomegalovirus (CMV) Reactivation After Allogeneic Stem Cell Transplantation
Brief Title: Autologous Cytomegalovirus (CMV)-Specific Cytotoxic T Cells for Cytomegalovirus (CMV) Reactivation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Miltenyi Biotec B.V. & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0620; NCI-2014-02335 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; Blood And Marrow Transplantation; Hematological malignancies; Cytotoxic T cells; CTL; Cytomegalovirus; CMV; Allogeneic hematopoietic stem cell transplantation; HSCT
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs) (Experimental): CTL product given as single infusion within 72 hours of CMV reactivation. CTL dose infused will be at a maximum dose of 10e5 viable CD3+ T cells/kg.
  Interventions: Biological: Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs)

INTERVENTIONS:
Biological: Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs) — CTL product given as single infusion within 72 hours of CMV reactivation. CTL dose infused will be at a maximum dose of 10e5 viable CD3+ T cells/kg.

SUMMARY:
The goal of this clinical research study is to learn if giving cytotoxic T lymphocytes (CTLs) can help control CMV when it reactivates (becomes active again) in patients who receive an allogeneic stem cell transplant. Researchers also want to learn about the safety of giving CTLs to patients who have had a stem cell transplant.

DETAILED DESCRIPTION:
The CTLs:

Blood (about 34 tablespoons) will be drawn 1 time. The blood will be frozen and stored in a laboratory at MD Anderson for future use to make the CTLs. If CMV comes back after your transplant, the blood will be used to create CTLs. To create CTLs, blood cells are grown in the laboratory and trained to kill CMV. If the blood is not used to make the CTLs within 3 years, it will be destroyed.

CTL Administration:

If your CMV becomes active after your stem cell transplant, you will receive the CTLs through a needle in your vein over 1-5 minutes one time, within 72 hours after CMV becomes active again. Before you receive the CTLs, you will receive Benadryl (diphenhydramine) and Tylenol (acetaminophen) by mouth to help reduce the risk of side effects. This can be done in either the hospital (if not yet discharged after your transplant) or in the outpatient clinic (if you are discharged).

Your vital signs will be monitored at the end of the infusion, and then at 30 and 60 minutes after the infusion. Your oxygen level will be measured by pulse oximetry. For this test, a clothespin-shaped clip will be placed on your finger for at least 30 minutes. If you are an outpatient, you will remain in the clinic for at least 1 hour after the CTL infusion.

If the CMV does not become active again after your stem cell transplant, you will not receive the CTL infusion.

Study Visits:

If the CMV does not become active again after your stem cell transplant, you will not receive the CTL infusion and your follow-up care will be done as per post-transplant standard of care.

If you receive the CTL infusion, you will have the tests/procedures listed below.

Within 48 hours before the CTL infusion:

* You will have a physical exam.
* Blood (about 6 tablespoons) will be drawn for routine tests and to check your kidney and liver function. Part of blood draw will be used for a pregnancy test for women who are able to become pregnant. To take part in this study, you must not be pregnant.

Once a week for 4 weeks, blood (about 4-8 tablespoons) will be drawn to check the level of CMV infection in your body. This may be done more often, if you doctor thinks it is needed.

About 1, 2, 3, and 4 weeks, and then about 3, 6, and 12 months after the CTL infusion:

* You will have a physical exam.
* Blood (about 4 tablespoons) will be drawn for routine tests and to check your kidney and liver function.

Blood (about 4 tablespoons) will be drawn for tests to learn more about the way the CTLs are working and how long they last in the body. This blood will be drawn before the CTL infusion, and then about 2 weeks, 4 weeks, 3 months, and 6 months after the CTL infusion. If possible, the blood needed for these tests will be collected during blood draws for routine tests so that no additional needle sticks will be needed.

Follow-Up Visits:

Once a week for 6 weeks, and then about 3, 6, 9, and 12 months after the CTL infusion, you will be checked for signs of graft-versus-host disease (GVHD) at every clinic visit. You were told about GVHD at the time of being prepared for transplant.

Length of Study:

Your participation on this study will end after your last follow-up visit about 12 months after the CTL infusion.

This is an investigational study. The use of CTLs to treat CMV infection is not FDA approved. At this time, CTLs are only being used to treat infections in research studies.

Up to 105 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. STEP 1: Within 30 days of study entry: Patients with a history of bone marrow disorders including hematological malignancies and aplastic anemia, Myelodysplastic Syndrome (MDS) and Myeloproliferative disorder (MPD) planning to undergo allogeneic HSCT with reduced intensity or myeloablative conditioning regimens.
2. Disease status must be complete remission by standard criteria for Lymphoma and Acute Leukemia patients.
3. Patients with Myelodysplastic Syndrome (MDS) and Myeloproliferative Disorder (MPD) must have <5% blasts in the bone marrow.
4. Patients with T Cell ALL must be in complete remission and MRD negative (-) by flow cytometry and molecular studies.
5. Patients >/= 18 years of age.
6. Karnofsky greater than or equal to 80%.
7. CMV seropositive.
8. Donor is either matched related, matched unrelated, mismatched unrelated, or haploidentical. Cord blood recipients are also eligible.
9. Hgb greater than 10 g/L.
10. Patient or patient's legal representative, parent(s) or guardian able to provide written informed consent.
11. Negative pregnancy test in female patients of childbearing potential.
12. STEP 2: Eligibility at time of generating and infusing CMV-specific cytotoxic T cells (adoptive immunotherapy): CMV reactivation defined as CMV DNAemia >/= 137 copies/ml.
13. Evidence of neutrophil engraftment defined as the absolute neutrophil count (ANC)> 0.5 X 10^3/for 3 consecutive days.
14. Clinical status to allow tapering of steroids to less than 0.5 mg/kg/day prednisone or equivalent.
15. Negative pregnancy test in female patients of childbearing potential.

Exclusion Criteria:

1. STEP 1: Within 30 days of study entry: T cell leukemia or lymphoma.
2. CMV seronegative.
3. Positive for HIV, HBV, HCV, HTLV1 and/or HTLV2.
4. STEP 2: Eligibility at time of generating and infusing CMV-specific cytotoxic T cells (adoptive immunotherapy): Documented CMV end-organ disease.
5. Patients receiving ATG, or Campath within 28 days of CMV reactivation.
6. Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to generating CTLs. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to generating CTLs. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
7. Patients who have received donor lymphocyte infusion (DLI) within 28 days.
8. Patients with active acute GVHD grades II-IV.
9. Active and uncontrolled relapse of malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betul Oran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in UT MD Anderson Cancer Center.
Pre-assignment Details: Five participants did not receive treatment as either they did not have CMV reactivation or had relapse of their primary malignancy and received treatment for relapse.
Period: Overall Study
Arm/Group | Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-Relapse Mortality
Description: Non-relapse mortality defined as death because of causes other than relapse of the underlying hematological malignancy.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs)
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Success Rate of Cytotoxic T Cells
Description: Treatment considered a success if the patient does not require initiation of cytomegalovirus (CMV) anti-viral therapy.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs)
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Cytomegalovirus (CMV)-Specific Cytotoxic T Cells (CTLs)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT02210065/Prot_SAP_000.pdf